CLINICAL TRIAL: NCT05404425
Title: Non-severe Traumatic Injuries Evaluation Using smartPhone Camera for Extra-hospital Regulation
Acronym: NIEPCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NIEPCE Trial
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Mild Traumatic Injury; Pre-hospital Dispatching; Visioconference

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visioconference: live visual injury evaluation (Experimental): For patients randomized in the intervention group, a live visual evaluation of the injury is performed by the Emergency Medical Call Center physician using a dedicated, secure smartphone app
  Interventions: Procedure: Visioconference: live visual injury evaluation
- Standard Procedure (Other): Usual management of patients
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Visioconference: live visual injury evaluation — For patients randomized in the intervention group, a live visual evaluation of the injury is performed by the Emergency Medical Call Center physician using a dedicated, secure smartphone app
  Arms: Visioconference: live visual injury evaluation
Procedure: Control — For patients randomized in the control group, the evaluation is performed by the Emergency Medical Call Center physician only by pone call
  Arms: Standard Procedure

SUMMARY:
Photography teletransmission allow a better and optimized dispatching of patients calling an Emergency Medical Call Center (EMCC) for a mild traumatic injury. It has previously been studied for patients to whom an ambulance was sent and therefore presumed to be older or with co-morbidities. The present trial aim to evaluate in the general population, the effect of a smartphone-mediated visioconference in the dispatching of patients calling an EMCC for mild traumatic injury.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years of age),
* free of will (not under any guardianship or liberty privation),
* suffering from Mild Traumatic Injury,
* availability of a smartphone with internet connection for the patients or witness,
* consenting to participate in the study

Exclusion Criteria:

* severe trauma requiring immediate medical assistance
* trauma associated with head injury, on antiplatelet therapy (APT) or anti-coagulation therapy (ACT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients dispatched elsewhere than to the nearest hospital | 1 year
  Proportion of patients dispatched elsewhere than to the nearest hospital (left at home for outpatient care / referred to a higher-level hospital / handled by MICA for advanced pre-hospital medical care)

SECONDARY OUTCOMES:
Under-triage | 1 year
  Under-triage : the proportion of patients initially left at home for outpatient care who had to visit an ED within the 10 following days for care related to the initial traumatic injury
Over-triage | 1 year
  Over-triage : the proportion of patients initially dispatched to an ED who could have underwent outpatient care

CONTACTS AND LOCATIONS:
Locations (1):
- Chu of Poitiers, Poitiers, France